CLINICAL TRIAL: NCT01862380
Title: Evaluation of Adrenocortical Functions by Insulin Tolerance Test and Sodium Depletion in Women With Nonclassical Congenital Adrenal Hyperplasia Due to 21-hydroxylase Deficiency in Comparison With Healthy Volunteers.
Brief Title: Adrenocortical Functions in Women With Nonclassical 21-hydroxylase Deficiency.
Acronym: EVAF-21
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P111005
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Adrenal Hyperplasia, Congenital; 21-hydroxylase Deficiency
Keywords: Adrenocortical function; Adrenal hyperplasia, Congenital; 21-hydroxylase; deficiency; cortisol; replacement therapy; Woman; Healthy people
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cases (Experimental): Functional explorations of cortisol and aldosterone production during stimulation by ITT and sodium depletion respectively in female patients with non classical 21-hydroxylase deficiency.
  Interventions: Other: Functional explorations
- Control (Experimental): Functional explorations of cortisol and aldosterone production during stimulation by ITT and sodium depletion respectively in healthy female controls.
  Interventions: Other: Functional explorations

INTERVENTIONS:
Other: Functional explorations — Functional explorations of cortisol and aldosterone production during stimulation by ITT and sodium depletion respectively
  Arms: Cases
Other: Functional explorations — Functional explorations of cortisol and aldosterone production during stimulation by ITT and sodium depletion respectively
  Arms: Control

SUMMARY:
The risk of adrenal insufficiency in patients with nonclassical congenital adrenal hyperplasia due to 21-hydroxylase deficiency is not well documented. Indication of cortisol replacement therapy in situation of acute stress or at long term is thus controversial. The mineralocorticoid reserve of these patients has never been evaluated.

Hypothesis: The glucocorticoid and mineralocorticoid function of the adrenal glands in women with nonclassical 21-hydroxylase deficiency is comparable with the adrenal functions of healthy age- sexe- and BMI-matched subjects.

DETAILED DESCRIPTION:
The primary end-point of the study is to evaluate the glucocorticoid function of the adrenal glands in women with nonclassical 21-hydroxylase deficiency (= patients) by comparing the maximal cortisol concentrations obtained during insulin tolerance test (ITT) in the patients and in the healthy volunteers.

The secondary end-point of the study is to determine the % of patients with a maximal plasma cortisol concentration greater or equal to 18μg/dL during ITT; compare the maximal plasma ACTH and salivary cortisol concentration during ITT in the two study groups; to evaluate the mineralocorticoid function of the patients by comparing the variations (changes from baseline) of the plasma renin, aldosterone, urinary aldosterone, systolic and diastolic blood pressure and pulse wave velocity in response to sodium depletion in the patients and in the healthy volunteers.

Women with nonclassical 21-hydroxylase deficiency followed in the Endocrinology and reproduction illnesses Service of the BICETRE Hospital, LE KREMLIN-BICETRE, France and female healthy volunteers will be proposed to participate.

Before inclusion patients must be genotyped and both patients and healthy volunteers must undergo an ACTH (Synacthen 250 μg IV) test for plasma cortisol and 17-hydroxyprogesterone concentration assessments.

After inclusion:

* ITT: IV injection of 0.10-0.2U/kg of insulin (ACTRAPID) at 09h00, dose adapted to BMI, with repeated measures 15, 30, 45, 60, 90 and 120 minutes after insulin injection for assessment of the glucocorticoid function, at the One Day Hospital of the Endocrinology and reproduction illnesses Service of the BICETRE Hospital, LE KREMLIN BICETRE.
* Sodium depletion test: obtained by PO administration of 40 mg of furosemide (LASILIX) at 09h00 in combination with low sodium diet (20mmol of Na/day) with repeated measures for assessment of the mineralocorticoid function during 24 hours after the drug administration at the Clinical Investigation Center of The George POMPIDOU Hospital, Paris.

ELIGIBILITY:
Inclusion Criteria:

Groupe of patients:

* women aged 18-50 years with nonclassical 21-hydroxylase deficiency with homozygous or compound heterozygous mutations of CYP21A2 and plasma 17-hydroxyprogesterone concentration after stimulation with synacthen >= 10ng/mL

Groupe of healthy volunteers :

* age matched female healthy volunteers with plasma 17-hydroxyprogesterone concentration after stimulation with synacthen < 2ng/mL

Exclusion Criteria:

* treatment with oral or local glucocorticoids < 1 year
* oral estroprogestative contraception < 3 months
* spironolactone < 3 months
* cyproterone acetate < 3 months
* treatment modifying the activity of the renin - angiotensine - aldosterone system < 2 weeks
* pregnancy and lactation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Maximal plasma cortisol concentration | Before and up to two hours after Insulin injection (Insulin tolerance test)
  Repeated measures 15, 30, 45, 60, 90 and 120 minutes after insulin IV injection

SECONDARY OUTCOMES:
% of patients with maximal plasma cortisol concentration >=18microg/dl | Before and up to two hours after Insulin injection (Insulin tolerance test)
  Repeated measures 15, 30, 45, 60, 90 and 120 minutes after insulin IV injection
Maximal plasma ACTH concentration | Before and up to two hours after Insulin injection (Insulin tolerance test)
  Repeated measures 15, 30, 45, 60, 90 and 120 minutes after insulin IV injection
Maximal salivary cortisol concentration | Before and up to two hours after Insulin injection (Insulin tolerance test)
  Repeated measures 15, 30, 45, 60, 90 and 120 minutes after insulin IV injection
Variation (change from baseline) of plasma rennin and plasma aldosterone concentration | Before and up to 24 hours after oral furosemide administration (Sodium depletion test)
  Repeated measures 1, 2, 3, 6, 9, 12, 24 hours after oral furosemide administration
Variation (change from baseline) of urinary aldosterone concentration | Before and up to 24 hours after oral furosemide administration (Sodium depletion test)
  Repeated measures in 4-hour urine portions after oral furosemide administration
Variation (change from baseline) of the systolic, diastolic blood pressure and pulse wave velocity | Before and up to 24 hours after oral furosemide administration (Sodium depletion test)
  Repeated measures 1, 2, 3, 6, 9, 12, 24 hours after oral furosemide administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kamenicky, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris - Bicêtre Hospital
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Bicêtre Hospital, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Kamenicky P, Blanchard A, Lamaziere A, Piedvache C, Donadille B, Duranteau L, Bry H, Gautier JF, Salenave S, Raffin-Sanson ML, Genc S, Pietri L, Christin-Maitre S, Thomas J, Lorthioir A, Azizi M, Chanson P, Le Bouc Y, Brailly-Tabard S, Young J. Cortisol and Aldosterone Responses to Hypoglycemia and Na Depletion in Women With Non-Classic 21-Hydroxylase Deficiency. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz005. doi: 10.1210/clinem/dgz005. PMID 31529070